Statistical analysis plan

# GEIS-30 STATISTICAL ANALYSIS PLAN

No EudraCT: 2012-002745-38

VERSION: V2.1 from November 29th, 2018



**TITLE:** Pazopanib phase II clinical trial to evaluate activity and tolerability in patients with advanced and / or metastatic liposarcoma who have relapsed to standard therapy or in those in whom there is no standard therapy.

#### **SPONSOR**

GRUPO ESPAÑOL DE INVESTIGACIÓN EN SARCOMAS, GEIS



1

Statistical analysis plan

# **COORDINATORS OF THE STUDY**

| COORDINATOR INVESTIGATOR GENERAL OF THE STUDY: |
|---------------------------------------------------|
| COORDINATOR INVESTIGATOR OF THE STUDY IN GERMANY: |
| COORDINATOR OF THE TRANSLATIONAL STUDY: |
| BEIS TECHNICAL SECRETARY: |

# Statistical analysis plan

# **INDEX**

| 1. | SUMMARY | 5 |
|---|---|---|
| 1.1. | SPONSOR OF THE STUDY | 5 |
| 1.2. | TITLE OF THE STUDY | 5 |
| 1.3. | PROTOCOL CODE | 5 |
| 1.4. | COORDINATING INVESTIGATORS | 5 |
| 1.4.1 | .COORDINATOR GENERAL COORDINATOR OF THE STUDY: | 5 |
| | .COORDINATOR OF THE STUDY IN GERMANY: | 5 |
| | COORDINATOR OF THE TRANSLATIONAL STUDY | 5<br>5<br>5<br>5<br>5 |
| | ETHICAL COMMITTEE OF CLINICAL RESEARCH THAT HAS APPROVED THE | |
| STU | DY | 5 |
| 1.6. | RESPONSIBLE MONITOR | 6 |
| 1.7. | STUDY TREATMENT | 6 |
| 1.8. | PHASE OF THE STUDY | 6 |
| 1.9. | MAIN OBJECTIVE OF THE STUDY | 6 |
| 1.10. | DESIGN | 6 |
| 1.11. | DISEASE OF STUDY | 6 |
| 1.12. | PRINCIPAL VARIABLE | 6 |
| 1.13. | STUDY POPULATION. NUMBER. TOTAL PATIENTS | 6 |
| 1.13. | 1. SAMPLE SIZE | 6 |
| 1.14. | DURATION OF THE TREATMENT | 6 |
| 1.15. | ESTIMATED CALENDAR OF THE STUDY | 6 |
| 1.16. | OBJECTIVES OF THE STUDY | 7 |
| 1.16. | 1. PRIMARY OBJECTIVE | 7 |
| 1.16. | 2. SECONDARY OBJECTIVES | 7 |
| | 3. TRANSLATIONAL OBJECTIVES | 7 |
| 1.16. | 4. POPULATIONS | 7 |
| 1.17. | GENERAL INCLUSION CRITERIA | 8 |
| | RESULTS | 11 |
| 2.1. | BASIC CHARACTERISTICS | 11 |
| 2.1.1 | SOCIODEMOGRAPHIC CHARACTERISTICS | 11 |
| 2.1.2 | .VITAL SIGNS | 12 |
| 2.1.3 | .HAEMATOLOGICAL PROFILE | 12 |
| 2.1.4 | .COAGULATION PROFILE | 12 |
| 2.1.5 | BIOCHEMICAL PROFILE | 12 |
| 2.1.6 | .THYROID FUNCTION | 13 |
| 2.1.7 | .URIANALYSIS | 14 |
| 2.1.8 | PREGNANCY TEST | 15 |
| 2.1.9 | .FUNCTIONAL STATUS: ECOG | 15 |
| 2.1.1 | 0. TUMOR CHARACTERISTICS AND PRE-TREATMENT LIPOSARCOMA | 16 |
| 2.1.1 | 0.1. INITIAL DIAGNOSIS | 16 |
| 2.1.1 | 0.2. RADIOTHERAPY | 18 |
| 2.1.1 | 0.2.1. RELAPSE AND TYPE OF TREATMENT | 18 |
| 2.1.1 | 0.3. PREVIOUS CHEMOTHERAPY | 19 |
| 2.1.1 | 1. PREVIOUS PATHOLOGY | 20 |
| 2.1.1 | 2. PHYSICAL EXAM | 21 |
| 2.2. | COMPLIANCE WITH TREATMENT VISITS | 23 |
| 2.3. | POPULATIONS ITT and PP | 24 |
| 2.4. | DURATION OF THE TREATMENT WITH PAZOPANIB | 24 |
| 2.5. | GLOBAL MONITORING | 25 |
| 2.6. | EFFICACY: MAIN ENDPOINT | 26 |
| 2.6.1 | EFFICACY BASED ON LOCAL ASSESSMENTS. ITT | 26 |
| 2.6.2 | EFFICACY BASED ON LOCAL ASSESSMENTS. PP | 26 |
| 2.6.3 | BASED ON CENTRALIZED ASSESSMENTS. ITT | 28 |

# Statistical analysis plan

| 2.6.4.EFFICACY BASED ON CENTRALIZED ASSESSMENTS. PP | 29 |
|----------------------------------------------------------------------|----|
| 2.7. EFFICACY: PROGRESSION FREE SURVIVAL SECONDARY ENDPOINT (PFS) | 30 |
| 2.7.1.PFS. LOCAL ASSESSMENT. ITT | 30 |
| 2.7.2.PFS. LOCAL ASSESSMENT. PP | 31 |
| 2.7.3.PFS. CENTRAL ASSESSMENT. ITT | 32 |
| 2.7.4.PFS. CENTRAL ASSESSMENT. PP | 33 |
| 2.8. EFFICACY: OVERALL SURVIVAL SECONDARY ENDPOINT (OG) | 35 |
| 2.8.1.OS. ITT | 35 |
| 2.8.2.OS. PP | 36 |
| 2.9. GMI: GROWTH MODULATION INDEX | 38 |
| 2.10. ECOG EVOLUTION | 39 |
| 2.11. SAFETY: AEs AND TOXICITIES | 39 |
| 3. ANNEX I: EFFICACY ACCORDING TO GMI | 44 |
| 3.1. MAIN ENDPOINT ACCORDING TO GMI | 44 |
| 3.1.1.RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. ITT | 44 |
| 3.1.2.RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. PP | 44 |
| 3.1.3. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. ITT. IN EACH | |
| COHORT | 44 |
| 3.1.4. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. PP. IN EACH | |
| COHORT | 45 |
| 3.2. ENDPOINT SECUNDARIO PFS ACCORDING TO GMI | 46 |
| 3.2.1.PFS ACCORDING TO GMI. LOCAL ASSESSMENT | 46 |
| 3.2.2.PFS ACCORDING TO GMI. LOCAL ASSESSMENT. IN COHORTE A | 46 |
| 3.2.3. PFS ACCORDING TO GMI. LOCAL ASSESSMENT. IN COHORT B | 47 |
| 3.3. SECONDARY ENDPOINT SG ACCORDING TO GMI | 48 |
| 3.3.1.OS ACCORDING TO GMI. | 48 |
| 3.3.2.OS ACCORDING TO GMI. IN COHORT TO | 49 |
| 3.3.3.OS ACCORDING TO GMI. IN COHORT B | 49 |
| 3.4. ECOG (BASAL) ACCORDING TO GMI | 51 |
| 3.4.1.ECOG BASAL ACCORDING TO GMI. ITT | 51 |
| 3.4.2.ECOG BASAL ACCORDING TO GMI. PP | 51 |
| 3.5. GRADE FNCLCC (BASAL) ACCORDING TO GMI | 51 |
| 3.5.1.GRADE FNCLCC BASAL ACCORDING TO GMI. ITT | 51 |
| 3.5.2.GRADE FNCLCC BASAL ACCORDING TO GMI. PP | 52 |
| 4. ANNEX II: LISTING OF ALL RELATED TOXICITIES | 52 |

Statistical analysis plan

#### 1. SUMMARY

#### 1.1. SPONSOR OF THE STUDY OF THE

GRUPO ESPAÑOL DE INVESTIGACIÓN EN SARCOMAS, GEIS



#### 1.2. TITLE OF THE STUDY

Pazopanib phase II clinical trial to evaluate activity and tolerability in patients with advanced and / or metastatic liposarcoma who have relapsed to standard therapy or in those in whom there is no standard therapy.

#### 1.3. CODE OF THE PROTOCOL

GEIS-30

N°EudraCT: 2012-002745-38

#### 1.4. COORDINATING INVESTIGATORS

1.4.1. Research General Coordinator of the study:



1.5. ETHICAL COMMITTEE OF CLINICAL INVESTIGATION THAT HAS APPROVED THE STUDY



Statistical analysis plan

#### 1.7. STUDY TREATMENT

Single arm of treatment with Pazopanib 800 mg (2x400mg or 4x200 mg) administered as single agent once a day.

#### 1.8. PHASE OF THE STUDY

Phase II study of two cohorts, open, non-randomized and multicenter with 11 participating centers in Spain and 5 in Germany. Patients will receive oral Pazopanib at a dose of 800mg once daily until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient, or decision of the investigator.

#### 1.9. MAIN OBJECTIVE OF THE STUDY

The primary objective of this study is to evaluate the activity of Pazopanib in patients with advanced and / or metastatic liposarcoma through progression-free survival (PFS) determined at 12 weeks after the start of treatment (according to RECIST criteria 1.1 and central radiological review).

#### 1.10. **DESIGN**

Phase II study of two cohorts, open, non-randomized and multicenter with 11 participating centers in Spain and 5 in Germany. To evaluate the activity and tolerability of pazopanib in patients with advanced and / or metastatic liposarcoma who have relapsed after standard treatment or for whom there is no established treatment.

The drug will be investigated separately in the following liposarcoma subtypes (cohorts):

- Well-differentiated liposarcoma / dedifferentiated liposarcoma (ALT-WD)
- Myxoid liposarcoma / round cell liposarcoma.

#### 1.11. DISEASE IN STUDY

Advanced and / or metastatic liposarcoma.

## 1.12. MAIN ASSESSMENT VARIABLE

The primary efficacy endpoint for this study is progression-free survival (PFS) determined 12 weeks after the start of treatment (according to RECIST 1.1 criteria and central radiological review).

#### 1.13. STUDY POPULATION. NUMBER. TOTAL PATIENTS

Patients with advanced or metastatic liposarcoma who have recurred after standard treatments or for whom there is no established treatment will be included.

#### **1.13.1.** Sample size

Estimation of 74 patients (Maximum of 37 patients in 2 different cohorts).

#### 1.14. DURATION OF TREATMENT

Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or decision of the investigator.

#### 1.15. ESTIMATED CALENDAR OF THE STUDY

Start date: Third quarter of 2012.

First visit of the first patient (PVPP): Fourth quarter of 2012.

Total duration of the recruitment period: 30 months.

First visit of the last patient (PVUP): Second guarter of 2015.

Follow-up period: 12 months. End of study date: March 2, 2018.

Statistical analysis plan

#### 1.16. OBJECTIVES OF THE STUDY

#### 1.16.1. Primary objective

The objective of this study is to evaluate the activity of Pazopanib in patients with advanced and / or metastatic liposarcoma by means of progression-free survival (PFS) determined after 12 weeks of treatment (according to the RECIST criteria v1.1 and central radiological revision).

#### 1.16.2. Secondary objectives:

- Median progression-free survival (median PFS).
- Objective tumor response [Complete confirmed response (CR) and partial response (PR) defined by RECIST 1.1].
- Time to start of response.
- Duration of response.
- Overall survival (OS).
- Clinical benefit rate (CBR).
- Growth modulation index (GMI).
- Security profile (according to CTCAE, version 4.0).

#### 1.16.3. Translational objectives

#### **PRIMARY OBJECTIVES:**

- To assess the influence of the tumor's angiogenic state on the response to Pazopanib.
- To assess the profile of serum cytokines as an indicator of response to Pazopanib.

#### **SECONDARY OBJECTIVES:**

- To assess the density of microvessels (DMV) and the pathways of p53, MDM2, PTEN, and VEGF / PDGF by immunohistochemistry, their correlation with prognosis, and their role as predictors of treatment with Pazopanib (response, PFS, and OS).
- Assess serum levels of various angiogenic factors / cytokines using Luminex XMAP Technology at baseline, after the first 3 weeks of treatment, at the time of maximum response and in tumor progression and its predictive value for survival and response to treatment: VEGF-A, PIGF-1, SDF-1 alpha (CXCL12), TNF alpha, IL-8, IL-6, PDGF-beta, HGF, E-Selectin, ICAM1, MMP-9 and FGFb.
- Analyze the presence of mutations in PIK3CA to demonstrate whether those liposarcomas with mutations in PIK3CA define a subgroup of patients with a different response to Pazopanib.

## 1.16.4. Populations

#### Population for efficacy.

- Analysis by Intention to Treat (ITT): Efficacy analyzes will be calculated on the population by intention to treat. All patients participating in the study will be included in the efficacy analysis.
- Analysis by Protocol (PP): Efficacy analyzes will be calculated on the per protocol population. All patients participating in the study and who have received at least 3 weeks of treatment with Pazopanib (without major protocol deviations) will be included in the efficacy analysis.

#### Population for security.

 Any patient included in the study who has received at least a single dose of study medication will be evaluable for toxicity analyzes.

#### Statistical analysis plan

#### 1.17. GENERAL INCLUSION CRITERIA

A subject will be considered eligible for inclusion in this study if they meet each and every one of the following criteria:

- 1. Subjects must give their informed consent before performing any of the study evaluations or procedures and must be willing to comply with the treatment and established monitoring.
- 2. Age ≥ 18 years.
- 3. Histological diagnosis of liposarcoma of intermediate or high grade of malignancy with metastatic or locally advanced disease. A paraffin-fixed tumor block and / or lamellae with representative sections stained with H / E (hematoxylin / eosin) must be available for its central pathological review and classification of tumors into 2 eligible subtypes:
  - Well-differentiated liposarcoma / Undifferentiated liposarcoma (ALT- WD)
  - Myxoid liposarcoma / Round cell liposarcoma.
- 4. Patients must present documented disease progression within 6 months prior to the patient's entry into the study.
- 5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
- 6. Measurable disease by RECIST criteria v1.1. There must be at least one measurable lesion located outside of a previously irradiated area. If the only measurable lesion is in a previously irradiated area, there should be documented progression after radiation therapy within 6 months prior to the patient's entry into the study.
- 7. The patient should not be considered a candidate for surgery or to receive radical radiotherapy. Eg Patients in whom surgery / radiotherapy cannot have a curative intention due to the extension of the disease. In the case of radiotherapy, it may be limited by previous irradiation on the same area.
- 8. The patient must have been considered a non-candidate for systemic chemotherapy or must have received at least one line of chemotherapy for metastatic or refractory disease. Up to a maximum of 3 previous lines are allowed for advanced / metastatic disease.

Eg patients not candidates for chemotherapy treatment:

- By age, concomitant pathology or negative of the patient.
- Patients who received anthracyclines in the adjuvant setting are generally not eligible to receive this drug as the first line for advanced disease.
- Monorenal patients or> 60 years are usually not good candidates for treatment with standard doses of ifosfamide.
- 9. Tumor tissue from all subjects is required for biomarker study before / during treatment with the study drug.
- 10. The patient must be able to swallow and retain the study medication.
- 11. Adequate organ and system function, as defined in Table 1.

#### Table 1. Definitions of adequate organic function.

#### Statistical analysis plan



- Subjects should not have received transfusions within 7 days prior to screening evaluation.
- Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
- Concomitant elevations of bilirubin and AST / ALT above 1.0 x ULN are not allowed.
- If UPC ≥ 1, a 24-hour urine protein determination should be performed.
   Subjects must have a value <1 g to be eligible. The use of urinary dipstick is not allowed to assess basal kidney function.</li>
- 12. A woman is eligible to participate in this study if: She has no reproductive potential, which includes, in addition to pathological situations of infertility:
  - Hysterectomized patients.
  - Patients with bilateral oophorectomy.
  - Patients with bilateral tubal ligation.
  - Post-menopausal patients.

Women who do not use hormone replacement therapy must have had a complete cessation of menstruation for a period  $\geq$  1 year and be over 45 years old, OR, in some cases, have FHS levels> 40 mIU / mL and estradiol levels < 40pg / mL (<140 pmol / L). Women using hormone replacement therapy must have experienced a complete cessation of menstruation for a period of  $\geq$  1 year and be older than 45 years OR have documented evidence of menopause due to hormonal values of FSH and estradiol prior

In the case of fertile women, those patients who have a negative result of a serum pregnancy test during the 2 weeks prior to the first dose of the study drug (preferably as close to the first dose of the drug as possible) are eligible if they agree to use appropriate contraceptive measures. The appropriate methods (when used continuously and according to the instructions of the doctor and the product) are the following:

- Complete sexual abstinence that will begin during the 14 days prior to the first exposure to the study drug, will be continued throughout treatment within the clinical trial and will continue until at least 21 days after the last dose of the drug.
- Oral contraceptives, both progestins as monotherapy and in combination with other agents.
- Injectable progesterone.

to initiation of hormonal treatment.

#### Statistical analysis plan

- Levonorgestrel implants.
- Vaginal ring with estrogens.
- Percutaneous contraceptive patches.
- Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year.
- Sterilized male partner (vasectomy with documented azoospermia) prior to the entry of their partner into the study (provided they are a monogamous partner).
- Double barrier method: Male condom and cervical diaphragm / cap with vaginal spermicidal agent (foam / gel / film / cream / suppository).
- Breastfeeding women should discontinue the natural feeding of the baby before receiving the first dose of the study drug until 14 days after the last dose of treatment.
- 13. Left ventricular ejection fraction (LVEF) above the lower limit of normal for the institution, either by echocardiogram or MUGA.

Statistical analysis plan

#### 2. EXPECTED RESULT ANALYSIS

These table summarize the expected results analysis of the clinical trial using ITT (Intent to Treat), PP (Per Protocol) populations for efficacy analysis, and those patients evaluable for toxicity for safety analyzes. This report will include complete patient follow up through the end of the estudy.

Table 2. Patients evaluable for the study according to cohort

| | Cohort A | Cohort B | Total |
|----------|----------|----------|-------|
| Hospital | N (%) | N (%) | N (%) |
| Total | | | |

#### 2.1. BASAL CHARACTERISTICS Baseline

Characteristics will be presented for all evaluable patients, globally and according to each cohort

## 2.1.1. SOCIODEMOGRAPHIC CHARACTERISTICS

The proportion of men / women.

| | | Table 3. Sex | | |
|---------|----------|--------------|-------|--------------|
| | Cohort A | Cohort B | Total | p-value |
| Sex | N (%) | N (%) | N (%) | |
| Male | • | | | <del>_</del> |
| Female | • | • | | <del>_</del> |
| Total | | | | _ |
| 4. 01-1 | | | | |

<sup>1:</sup> Chi-square test

## Mean age.

Table 4. Age

| | | | | | Tubic T | - Agc | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cohort A | | | Co | hort B | Total | | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| Age | | | • | | · | | | | | |

<sup>1:</sup> Test Mann-Whitney U

#### 2.1.2. VITAL SIGNS

Statistical analysis plan

Table 5. Vital Signs

| | | | | | ,,, o | ai Oigiio | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cohort A | | | Cohort B | | | Total | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>( Min-Max) | - p-<br>value <sup>1</sup> |
| Height | | | | | | - | · | | | |
| Weight | | | | | | | | | | |
| BP Systolic | ; | | | | | | | | | |
| BP | | | | | | | | | | |
| Diastolic | | | | | | | | | | |
| Body | | | | | | | | | | |
| temperature | е | | | | | | | | | |
| 1: Mann Whit | 2011 | Litoot | | | | | | • | · | |

<sup>1:</sup> Mann-Whitney U test

## 2.1.3. HAEMATOLOGICAL PROFILE

Table 6. Haematological profile

| | | | i abic o | | Ciliatolo | gicai promic | • | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cohort A | | | Col | nort B | | Т | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean (<br>SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| Hemoglobin | | | | | | - | | | - | |
| Platelets | | | | | | | | | | |
| Neutrophils | | | | | | | | | | |
| Lymphocytes | 3 | | | | | | | | | |
| 4 5 4 3 5 4 11 | | | | | | • | | | | |

<sup>1:</sup> Mann-Whitney U test

#### 2.1.4. COAGULATION PROFILE

Table 7. Coagulation profile

| | | | | | р. о | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Cohort A | | | Co | hort B | | To | | |
| N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| Prothrombin | | | | | - | | | | |
| INR | | | | | | | | | |
| PTT | | | | | | | | | |
| 1. Mann Whitney | LLToot | | | | | | | | |

<sup>1:</sup> Mann-Whitney U Test

## 2.1.5. BIOCHEMICAL PROFILE

Table 8. Biochemical profile

| | | Co | hort A | | Cohort B | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Medi ana<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| Protein | | | • | | | | | | | |
| Albumin | | | | | | | | | | |
| BUN | | | | | | | | | | |
| Creatinine | | | | | | | | | | |
| Clearance | | | | | | | | | | |
| SGOT / AST | | | | | | | | | | |
| SGTP / ALT | | | | | | | | | | |
| Alkaline | | | | | | | | | | |
| Phosphatase | | | | | | | | | | |
| Bilirubin | | • | | | • | | | | | |

# Statistical analysis plan

| Phosphorus |
|------------------|
| Sodium |
| Potassium |
| Calcium |
| Chloride |
| Magnesium |
| Amylase |
| Lipase |
| Lactate |
| dehydrogenase |
| 4 84 18414 114 4 |

<sup>1:</sup> Mann-Whitney U test

# 2.1.6. THYROID FUNCTION

Table 9. Thyroid function

| Table 9. Thyroid function | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort A | | | | Cohort B | | | To | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| TSH | | • | • | | • | | | | • | |
| T4 | | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

#### Statistical analysis plan

#### 2.1.7. URIANALYSIS

Table 10. Urinalysis

| | Tabl | e io. Offically. | , i j | | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | p-value |
| | | N (%) | N (%) | N (%) | |
| | Normal | | | | |
| Dipstick Protein | Abnormal | | | | |
| | Not applicable | | • | | |
| | Total | | • | | |
| | Normal | | | | |
| Microscopic | Abnormal | | • | | |
| analysis | Not applicable | | | | |
| | Total | | | | |
| | Normal | | | | |
| 24-Hour | Abnormal | | | | |
| proteinuria | Not applicable | | | | <del></del> |
| | Total | | | | <del></del> |
| 4.4 | Ohi anuana O. Fiahanla ava | -4.44 | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

**Table 11. Urinalysis results** 

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | |
| | Normal / No result | | • | | |
| | (+) | | | | |
| | 0.25 | | | | |
| <b>5</b> " | 1+ | | • | | _ |
| Result | 13 | | • | | |
| Dipstick<br>Protein | 14 | | | | |
| Protein | 25 mg / dl | | • | | |
| | negative | | • | | _ |
| | traces | | • | | |
| | Total | | | | |
| Abnormal | Normal / No result | | | | |
| microscopic | Erythrocyts | | • | | |
| analysis <sup>.</sup> | Total | | • | | |
| | 4 01: 0 5:1 1 | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Table 12. 24-hour proteinuria

| | | Cohort A | | | Co | hort B | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| 24-Hour | | | • | | • | • | | | • | |
| Result | | | | | | | | | | |
| proteinuria | | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U Test

#### 2.1.8. PREGNANCY TEST

Table 13. Pregnancy test

## Statistical analysis plan

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | _ | N (%) | N (%) | N (%) | • |
| Pregnancy<br>test) | Negative | | | | |
| | Total | | | | _ |
| Turns of Took | Serum | | , | | |
| Type of Test | Total | | , | | _ |
| | 1: Chi-square test | | | | |

Table 14. Test details of pregnancy

| Patient | Cohort | Sex | Age | Pregnancy<br>test | Type of<br>pregnancy<br>test | Reason test not performed |
|---|---|---|---|---|---|---|

# 2.1.9. FUNCTIONAL STATUS: ECOG

Table 15. ECOG at baseline

| | | | Iab | ie io | . ECUG | at baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ECOG at | | Coho | rt A | | Coho | ort B | | То | tal | |
| baseline | | N ( | %) | | N ( | %) | | N (%) | | p-<br>value <sup>1</sup> |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | _ |
| Total | | | | | | | | | | <b>=</b><br> |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | p-<br>value <sup>3</sup> |
| Baseline<br>ECOG | | | | | | | | | | · |

<sup>1:</sup> Chi-square; 2: Fisher's exact test; 3: Test Mann-Whitney

Statistical analysis plan

# 2.1.10. TUMOR CHARACTERISTICS AND PRETREATMENT LIPOSARCOMA

2.1.10.1. Initial diagnosis

Table 16. Location of the tumor

| | | Cohort A | Cohort B | Total | p-value |
|-------------|-------------------|----------|----------|-------|--------------|
| | | N (%) | N (%) | N (%) | |
| | pelvic girdle | | | | |
| | Upper Limbs | • | , | | _ |
| Location of | Lower extremities | | | | |
| the tumor | Retro-peritoneum | • | , | | _ |
| | Others | • | | | <del>_</del> |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisherexact test

#### Other locations:

Table 17. Other tumor locations

| Table 111 Carlot tarrier locations | | |
|---|---|---|
| Patient | Cohort | Other locations |
| | <u>-</u> | · |

Table 18. Histological type (local review)

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | |
| | Well-differentiated<br>Liposarcoma | , , | . , | • • • | _ |
| Histological | Undifferentiated | | | | |
| type | Pleomorphic | | , | | |
| _ | Myxoid | | , | | <del></del> |
| - | Total | | | | |
| | 4 OL: 0 E: 1 I | | | • | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Histological diagnosis was also analyzed centrally.

Table 19. Histological type (centralized review)

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | |
| • | Liposarcoma distinct | | | | |
| Histological | well differentiated liposarcoma / dedifferentiated | | | | _ |
| type | liposarcoma undifferentiated | <u>.</u> | • | | = |
| (centralized) | liposarcoma myxoid | • | • | | <del>_</del> |
| · | Total | | | | _ |
| | 4. Chi. assussa O. Taat Fishassusst | | | | |

<sup>1:</sup> Chi -square; 2: Test Fisherexact

## comparison:

#### Statistical analysis plan

Table 20. GradeFNCLCC

| | | | Table 20. | Orauei | 10L00 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| GradeFNCLCC | | Coh | ort A | Coh | ort B | | То | tal | |
| • | | N ( | %) | N ( | (%) | | N ( | (%) | p-<br>value <sup>3</sup> |
| 1 | | | | | | | | | |
| 2 | | | | | | | | | _ |
| 3 | | | | | | | | | <b>=</b> ' |
| Total | | | | | | | | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max ) | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | p-<br>value <sup>3</sup> |
| Degree<br>FNCLCC | | - | · | • | | | • | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test; 3: Mann-Whitney U test

#### Previous treatments:

Table 21. Initial treatment

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | |
| Radiotherap | Yes | | | | _ |
| y for primary_<br>tumor | No | • | • | | |
| | Total | | | | |
| Initial<br>treatment | Yes | | | | _ |
| | No | • | • | | |
| | Total | | | | |
| | Radical surgery | - | | | |
| -<br>- | Wide | | | | |
| Type of | Marginal positive resection | • | • | | |
| initial<br>treatment - | Only biopsy | - | | | |
| | Others | | | | |
| | Total | | | | _ |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

## Other initial treatments:

Table 22. Other initial treatments

| Table 22. Other initial freatheries | | |
|-------------------------------------|--------|-------------|
| Patient | Cohort | Other types |

Elapsed time between initial treatment and Pazopanib treatment:

Table 23. Time from initial treatment to start of Pazopanib (years)

| | . u. | <del>510 </del> | | | · tioutiii | one to otal t or | | opailio ( | you.o, | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cohort A | | | Cohort B | | | To | | |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | - p-<br>value <sup>1</sup> |
| Time from | | | | | | | | | | |
| initial tt to | | | | | | | | | | |
| Pazopanib | | | | | | | | | | |

<sup>1:</sup> Mann U-test Whitney

Statistical analysis plan

#### 2.1.10.2. RADIOTHERAPY

Table 24. Radiotherapy

| | · | <u> </u> | - ti.io.upy | | |
|--------------|-------|----------|-------------|-------|-------------|
| | | Cohort A | Cohort B | Total | p-value |
| | _ | N (%) | N (%) | N (%) | |
| · | Yes | | • | | |
| Radiotherapy | No | | • | | <del></del> |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Elapsed time between initial treatment and Pazopanib treatment:

Table 25. Duration of radiotherapy (months)

| | | | Table 23. De | ura | tion of i | aulotherapy (i | IIOII | 1113 <i>)</i> | | |
|---|---|---|---|---|---|---|---|---|---|---|
| • | | Coh | ort A | | Co | hort B | | To | otal | - n |
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | medium<br>(Min-Max) | N | Mean<br>(SD) | median<br>(min-max) | - p-<br>value <sup>1</sup> |
| Duration of radiotherapy (months) | 1 | | | | | | | | | |

<sup>1:</sup> Test Mann-Whitney

# 2.1.10.2.1. RELAPSE and type of treatment

Table 26. Relapses and type of treatment

| | | Cohort a | Cohort B | Total | p-value |
|-----------------|-------|----------|----------|-------|-------------|
| | | N (%) | N (%) | N (%) | |
| | No | | | | |
| relapse | Yes | | , | | <del></del> |
| _ | Total | • | • | | |
| | No | | | | • |
| Metastasis | Yes | • | • | | |
| | Total | | | | |
| | No | • | • | | |
| Local relapse | Yes | | | | |
| | Total | • | • | | |
| | No | • | • | | |
| Other relapse | Yes | • | • | | |
| _ | Total | | | | |
| | No | • | • | | |
| radical surgery | Yes | • | | | |
| _ | Total | | | | |
| | No | • | • | | |
| wide Resection | Yes | • | • | | |
| | Total | | | | |
| Positive | No | | | | |
| marginal | Yes | | | | |
| resection | Total | | | | |
| Only biopsy | No | | | | |

#### Statistical analysis plan

| | Yes |
|------------------|-------|
| | Total |
| Other treatments | No |
| | Yes |
| | Total |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

#### 2.1.10.3. PREVIOUS CHEMOTHERAPY

Table 27. Previous chemotherapy

| | iubi | C 27. 1 1CVIOUS C | memoriapy | | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | — p-value |
| | | N (%) | N (%) | N (%) | — p-value |
| Danish | No | • | | | |
| Previous<br>chemotherapy | Yes | • | | | |
| | Total | • | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

The following table will include all the chemotherapy lines prior to Pazopanib. Patients could have received more than one line of chemotherapy.

Table 28. Prior Chemotherapy:List of treatments

| Prior Chemotherapy | Cohort A | Cohort B | Total |
|----------------------------------|----------|----------|-------|
| | N (%) | N (%) | N (%) |
| Adriamicine-Ifosfamide / 21 days | | | |
| Adriamicine | | | |
| Adriamicine / Ifosfamide / D | | | |
| actinomycin | | | |
| CCGM Phase I | | | |
| Cisplatin / Doxorubicin | | | |
| Dacarbazine | | | |
| Dacarbazine /Gemcitabin | | | |
| Docetaxel | | | |
| Docetaxel/ Gemcitabin | | | |
| Doxorubicin | | | |
| Epirubicin | | | |
| Eribulin | | | |
| Gemcitabin | | | |
| Gemcitabin / Taxotere | | | |
| lfosfamide | | | |
| Mesna Ifosfamide + | | | |
| Ifosfamide / ADRIBLASTIN + G-CSF | | | |
| lxoten | | | |
| Nilotinib | | | |
| p53-HDM2inhibitor interaction | | | |
| Tegafur | | | |
| TH-302 | | | |
| Trabectedin | | | |

Best initial response to chemotherapy:

#### Statistical analysis plan

prior chemotherapy Table 29.

| | | Cohort A | Cohort B | Total | n voluo |
|---|---|---|---|---|---|
| | - | N (%) | N (%) | N (%) | — p-value |
| Best previous — | CR | | | | |
| | PR | | | | |
| | SD | | • | | |
| | PD | | • | | |
| response - | WITHOUT | | | | |
| _ | ASSESSMENT | | | | |
| | Total | | | | |
| Relapse in _<br>last previous<br>chemotherapy | No | | | | |
| | Yes | | | | |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Global number of cycles and duration of initial chemotherapy:

Table 30. Number of cycles and duration of previous chemotherapy

| | | Cohort A | | | Coh | ort B | | To | otal | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-<br>Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | p-<br>value <sup>1</sup> |
| Total number of chemotherapy cycles | | | | | | | | | | |
| Duration of previous chemotherapy, until relapse (prior to Pazopanib) (days) | | | | | | | | | | |
| Time from previous relapse to start with Pazopanib (days)PREVIOUS | | | | | | | | | | |

<sup>(</sup>days)PREVIOUS

1: Mann-Whitney U test

#### **2.1.11. PATHOLOGY**

Table 31. Previous pathologies

| | | Cohort A | Cohort B | Total | p-value |
|---------------|-------|----------|----------|-------|---------|
| | | N (%) | N (%) | N (%) | |
| | No | | | | |
| Previous — | Yes | | • | | |
| pathologies — | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

The following table will include all pathologies prior to the start of treatment with Pazopanib. The patients could have presented more than one pathology.

#### Statistical analysis plan

Table 32. List of previous pathologies Previous

| pathologies | Cohort A | Cohort B | Total |
|-------------|----------|----------|-------|
| | N (%) | N (%) | N (%) |
| _ | | | |

#### 2.1.12. PHYSICAL EXAMINATION

Table 33. Physical exam

| | | Cohort A | Cohort B | Total | p-value |
|------------------|----------------|----------|----------|-------|---------|
| | _ | N (%) | N (%) | N (%) | |
| Cardiovascular | Normal | | | | |
| Carulovasculai | Total | | | | |
| Respiratory | Normal | | | | |
| | Abnormal | | | | |
| | Total | | | | |
| CNS | Normal | | | | |
| | Not performed | | | | |
| | Not applicable | | | | |
| | Total | | | | |
| | Normal | | | | |
| Gastrointestinal | Abnormal | | | | |
| | Total | | | | |
| | Normal | | | | |
| Musculoskeletal | Abnormal | | | | |
| Wiusculoskeletai | Not performed | | | | |
| | Total | | | | |
| | Normal | | | | |
| Dormatological | Abnormal | · | | · | |
| Dermatological | Not performed | | | | |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

The list of patients with abnormal results on the physical examination will be presented in the following table:

Table 34. Patients with abnormal results

# Statistical analysis plan

| Patient | Cohort | Examination | Result | Specify |
|---------|--------|-------------|--------|---------|

Statistical analysis plan

# 2.2. COMPLIANCE WITH TREATMENT VISITS

The status of completion of visits at the time of database lock:

**Table 35. Completion of treatment visits** 

| | | Cohort A | Cohort B | Total | p-value |
|------------------------|-------|----------|----------|-------|-------------|
| | | N (%) | N (%) | N (%) | |
| Baseline visit | Yes | | | | |
| completed | Total | | • | | |
| Vioit day 1 | No | | • | | |
| Visit day 1 completed | Yes | | | | |
| Completed | Total | | • | | |
| Visit week 1 | No | | | | |
| completed - | Yes | | | | |
| Completed | Total | | | | |
| Visit week 3 completed | No | | | | |
| | Yes | | | | |
| | Total | | | | |
| Visit week 5 | No | | • | | |
| completed – | Yes | | | | |
| Completed | Total | | | | |
| Visit week 7 | Yes | | • | | |
| completed | Total | | | | |
| Visit week 9 | No | | | | |
| completed - | Yes | | | | |
| Completed | Total | | | | |
| Visit week 12 | No | | • | | |
| completed - | Yes | | • | | |
| Completed | Total | | • | | |
| Complete completion | No | | · | | |
| from baseline to | Yes | | | | |
| week 12) | Total | | | | <del></del> |

1: Chi-square; 2: Fisher's exact test

Statistical analysis plan

#### 2.3. ITT and PP POPULATIONS

To determine ITT and PP populations, the definitions specified in the protocol will be followed:

- Analysis by Intention to Treat (ITT): Efficacy analyses will be calculated on the population by intention to treat. All patients participating in the study will be included in the efficacy analysis.
- Analysis by Protocol (PP): Efficacy analyzes will be calculated on the protocol population. All patients participating in the study and who have received at least 3 weeks of treatment with Pazopanib (without major protocol deviations) will be included in the efficacy analysis.

**Table 36. ITT and PP Populations** 

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | |
| ITT | Yes | | • | | |
| population | Total | | | | |
| | <3 weeks | | | | |
| Duration tt | ≥3 weeks | • | | | |
| Pazopanib (weeks) | Ongoing<br>(no end date of tt) | | | | |
| <del>-</del> | Total | | • | | |
| B l . (' | No | | • | | |
| Population - | Yes | | , | | <del></del> |
| PP - | Total | | | | |

<sup>1:</sup> Chi-square; 2: Test Fisherexact

Pacientes with less than 3 week of pazopanib treatment:

Table 37. Patients with duration of pazopanib <3 weeks

| Study Subject<br>ID | Cohort | PP<br>population | Reason excluded from PP population | Tx Pazopanib<br>duration (days) |
|---|---|---|---|---|

# 2.4. Duration of pazopanib

Table 38. Duration of Pazopanib treatment (days)

| | Cohort A | | Coh | Cohort B | | Total | | |
|---|---|---|---|---|---|---|---|---|
| | N Mean (SD) | Median<br>(Min-Max) | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min -Max) | value |
| Duration of treatment with Pazopanib <sup>2</sup> | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test; 2: For a patient that the end date of treatment with Pazopanib was not available, the date of PD / Exitus was taken as the end date of treatment.

Statistical analysis plan

# 2.5. GLOBAL FOLLOW-UP

Table 39. Global follow-up (weeks) ITT and PP

| | | Cohort A | | | Cohort B | | | T | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max)- | p-<br>value <sup>1</sup> |
| Global<br>follow-up<br>ITT | | | | • | | | | | | |
| Global<br>follow-up<br>PP | | | | | | | | | | |

<sup>1:</sup> Test Mann-Whitney

Statistical analysis plan

#### 2.6. EFFICACY: MAIN ENDPOINT

Following the instructions of the protocol primary efficacy endpoints in populations ITT and PP will be calculated following the criteria:

Patients who are alive and without evidence of progression at this time will be considered successes, and those who have progressed or died at this time will be considered treatment failures. Patients in whom progression is unknown or not available will also be considered failures. Diagnosis of progression should be based on measurements of tumor lesions, according to the RECIST 1.1 criteria.

#### 2.6.1. EFFICACY BASED ON LOCAL ASSESSMENTS. ITT

The tables below will analyze the **response at 6 and 12 weeks**, based on **local assessments** TAC.

Table 40. Response to treatment: Local assessments at 6 and 12 weeks ITT

| | | Cohort A | Cohort B | Total | n volue |
|---|---|---|---|---|---|
| | - | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | — p-value |
| Response | SD | | | , | |
| at | PD | | | | |
| 6 weeks | Total | | | | <del></del> |
| Response | SD | | | | <u> </u> |
| to | PD | | | · | |
| 12 weeks | Total | | | | <del></del> |

<sup>1:</sup> Chi-square; 2: Test exacto de Fisher

Responses will be recoded according to **clinical benefit (CR, RP or EE)** and in the ITT population, both at 6 and 12 weeks.

Table 41. Clinical benefit, response to treatment: Local assessments at 6 and 12 weeks ITT

| | | Cohort A | Cohort B | Total | n valua |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | — p-value |
| Response | Yes | | | | |
| at<br>6 weeks | No (PD) | | | | |
| CLINICAL<br>BENEFIT | Total | | | | _ |
| Response | Yes | | | | |
| at<br>12 weeks<br>CLINICAL<br>BENEFIT | No (PD) | | • | | |
| | Total | | | | _ |
| | | | | | _ |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

#### 2.6.2. EFFICACY BASED ON LOCAL ASSESSMENTS. PP

In the PP population, both at 6 and 12 weeks.

#### Statistical analysis plan

Table 42. Response to treatment: Local assessments at 6 and 12 weeks PP

| | | Cohort A | Cohort B | Total | _ p-value |
|---|---|---|---|---|---|
| | _ | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | — p-value |
| Response | SD | | | | |
| at | PD | | | | <del></del> |
| 6 weeks | Total | | | | <del></del> |
| Response | SD | | | | |
| to<br>12 weeks | PD | | | | <del></del> |
| | Total | | | | _ |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

The responses will be recoded according to the **clinical benefit (CR, RP or EE)** and in the PP population, both at 6 and 12 weeks.

Table 43. Clinical benefit, response to treatment: Local evaluations at 6 and 12 weeks PP

| | | Cohort A | Cohort B | Total | n volue |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | – p-value |
| Response | Yes | | | | |
| at<br>6 weeks | No (PD) | | | | |
| CLINICAL<br>BENEFIT | Total | | | | |
| Response | Yes | | | | |
| at<br>12 weeks | No (PD) | | | | |
| CLINICAL<br>BENEFIT | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

#### 2.6.3. BASED ON CENTRALIZED ASSESSMENTS. ITT

The tables below will record the **response at 6 and 12 weeks**, based on **centralized assessments** TAC. As for the local evaluations. The centralized evaluations will be reviewed following the criteria specified in the protocol for the evaluation of the main endpoint:

"Patients who are alive and without evidence of progression at this time will be considered as successes, and those who have progressed or died at this time will be considered as treatment failures. Patients in whom it is unknown whether or not there is progression will also be considered as failures."

In the ITT population, both 6 and 12 weeks.

Table 44. Response to treatment: Value. Centralized at 6 and 12 weeks ITT

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | _ | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | · |
| | PD | | | | |
| Response | SD | | | • | |
| at<br>6 weeks | PR | | | | |
| O WEEKS | Total | | | | |
| | PD | | | | |
| Response<br>at<br>12 weeks | SD | | | | |
| | PR | | | | <del></del> |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Responses will be recoded according to **clinical benefit (CR, RP or EE)** and in the ITT population.

Table 45. Clinical benefit, response to treatment: Value. centralized at 6 and 12 weeks ITT

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | <del>_</del> · |
| Response | Yes | | | | |
| at<br>6 weeks | No (PD ) | | | | <u> </u> |
| CLINICAL<br>BENEFIT | Total | | | | |
| Response | Yes | | | | |
| at<br>12 weeks | No (PD) | | | | _ |
| CLINICAL<br>BENEFIT | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

#### 2.6.4. EFFICACY BASED ON CENTRALIZED ASSESSMENTS. PP

Table 46. Response to treatment: Centralized evaluations at 6 and 12 weeks PP

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | _ | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | <u> </u> |
| | PD | | | | |
| Response | SD | | | | |
| at<br>6 weeks | PR | | | | |
| o weeks | Total | | • | • | |
| D | PD | | | | |
| Response | SD | | • | • | |
| at<br>12 weeks | PR | | • | • | |
| | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Responses will be recoded according to **clinical benefit (CR, RP or EE)** and in the PP population.

Table 47. Clinical benefit, response to treatment: Centralized evaluations at 6 and 12 weeks PP

| | | Cohort A | Cohort B | Total | p-value |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | _ ' |
| Response | Yes | | | | |
| at<br>6 weeks | No (PD) | | | | |
| CLINICAL<br>BENEFIT | Total | | | • | |
| Response | Yes | | | | |
| at<br>12 weeks | No (PD) | | | | <del></del> |
| CLINICAL<br>BENEFIT | Total | | | | |
| | | | | | _ |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

# 2.7. EFFICACY: SECONDARY ENDPOINT PROGRESSION FREE SURVIVAL (PFS)

#### 2.7.1. PFS. LOCAL ASSESSMENT. ITT

Table 48. Progression-free survival at 12 and 24 weeks according to cohorts (local

| | | ass | <u>essment</u> | . ITT) | | | |
|---|---|---|---|---|---|---|---|
| Progression-f | ree survival | N<br>events | N<br>patients<br>at risk | cumulativ | imated<br>ve survival<br>itio | 95% CI | |
| | Cohort | | | | | | |
| at 40 waalsa | Α | | | | | | |
| at 12 weeks — | Cohort | | | | | | |
| | В | | | | | | |
| | Cohort | | | | | | |
| ot 24 wooks — | Α | | | | | | |
| at 24 weeks — | Cohort | | • | • | - | | <del></del> |
| | В | | | | | | |
| | Strategy | N (%)<br>events | Median<br>(weeks) | Min-Max | Standard error | 95% CI | p-<br>value |
| Dua nua ani an | Α | | | | | | |
| Progression- free survival — | В | | | | | | |
| iree survival — | Total | | | | | | |
| | 1: Log-rank t | est | | | | | |

1: Log-rank test

Figure 1. Progression-free survival according to cohorts ( Local assessment ITT). Kaplan-Meier curve.

Table 49. Progression during follow-up (local assessment. ITT)

| | | Cohort A | Cohort B | Total | _ n_ |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%,<br>95% CI) | — p-<br>value |
| | PD | | | | |
| Progression-<br>free survival | Alive: Free of progression | | | | |
| | Total | · | · | · | |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

Table 50. Types of progressions / censorship during follow-up (local assessment. ITT)

| | | Cohort<br>A | Cohort<br>B | Total | · p-value |
|---|---|---|---|---|---|
| | | N (%,<br>95% CI) | N (%,<br>95% CI) | N (% ,<br>95% CI) | p-value |
| _ | Progression-Disease | | | | |
| | progression Clinical progression | | - | - | <del>-</del> |
| Progression- | Alive without PD at the end<br>of follow-up | - | - | - | |
| free survival | Alive without PD: censored<br>by surgery | _ | | | - |
| | Alive without PD:<br>abandonment due to<br>patient decision | | | | • |
| | Total | | | | - |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

#### Statistical analysis plan

Table 51. Time to PD (weeks) (Local assessment, ITT)

| | | Cohort A | | | Cohort B | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min- Max) | N | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |
| Time to PD<br>(weeks) | | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

## 2.7.2. PFS. LOCAL ASSESSMENT. PP

Table 52. Progression-free survival at 12 and 24 weeks according to cohorts (local assessment. PP)

| Progression | -free survival | N events | N patients at risk | | ed cumulative<br>ival ratio | 95% CI | |
|---|---|---|---|---|---|---|---|
| at 12 | Cohort A | | | | | | |
| weeks | Cohort B | | | | | | |
| at 24 | Cohort A | | | | | | |
| weeks | Cohort B | | | | | | |
| | Strategy | N (%)<br>events | Median<br>(weeks) | Min-Max | Standard error | 95% CI | p-value <sup>1</sup> |
| Progressi | Α | | | | | | |
| on-free | В | | | | | | |
| survival | Total | | | | | | |

<sup>1:</sup> Log-rank test

Figure 2. Progression-free survival according to cohorts ( Local assessment PP). Kaplan-Meier curve.

| | | Cohort A | Cohort B | Total | _ |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95%<br>CI) | – p-<br>value |
| _ | PD | | | | |
| Progressio —<br>n-free<br>survival — | Alive: Free of progression | | | | _ |
| | Total | | | | |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

Table 54. Types of progressions / censorship during follow-up (local. PP)

| | | Cohort A | Cohort B | Total | |
|---|---|---|---|---|---|
| | | N (%, 95% | N (%, 95% N | l (% , 95% | p-value |
| | | CI) | CI) | CI) | |
| | Progression-Disease | | | | |
| | progression Clinical progression | | | | = |
| Progressio | Alive without PD at the end of follow- | _ | · · | | - |
| n-free | up | | | | _ |
| survival | Alive without PD: censored by | | | | -" |
| | surgery | | | | |
| | Alive without PD: abandonment due to patient decision | _ | | | |

#### Statistical analysis plan

#### Total

1: Pearson Chi-square; 2: Fisher's exact test

Table 55. Time to PD (weeks) (Local. PP)

| | Cohort A | | | Cohort B | | | | Tot | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min- Max) | N | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |
| Time to PD (weeks) | | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

#### 2.7.3 PFS. CENTRAL ASSESSMENT. ITT

To describe the event in PFS, the protocol will be followed:

"Overall progression-free survival will be calculated from the date of initiation of treatment to the first date of documented progression or date of death, whatever the cause. Live patients with no evidence of progression at the time of analysis will be censored on the date of the last follow-up."

Table 56. Progression-free survival at 12 and 24 weeks according to cohorts (Central assessment. ITT)

| | | usse | 331110111 | <i>,</i> | | | |
|---|---|---|---|---|---|---|---|
| Progression-f | ree survival | N<br>events <sup>p</sup> | N<br>patients<br>at risk | cumulativ | imated<br>ve survival<br>itio | 95% CI | |
| | Cohort | | | | | | |
| at 12 weeks - | Α | | | | | | |
| | Cohort | | | | | | |
| | В | | | | | | |
| | Cohort | | | | | | |
| at 24 weeks — | Α | | | | | | |
| at 24 weeks — | Cohort | | • | | - | | |
| | В | | | | | | |
| | Strategy | N (%)<br>events ( | Median<br>(weeks) | Min-Max | Standard error | 95% CI | p-<br>value <sup>1</sup> |
| Dunananian | Α | | | | | | |
| Progression- | В | | | | | | |
| free survival — | Total | | | | | | _ |
| | 1. Log rank t | toet | | | | | |

<sup>1:</sup> Log-rank test

Figure 3. Progression-free survival according to cohorts ( Central assessment ITT). Kaplan-Meier curve.

#### Statistical analysis plan

Table 57. Progression during follow-up (Central assessment. ITT)

| | | Cohort A | Cohort B | Total | |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%,<br>95% CI) | – p-<br>value |
| | PD | | | | |
| Progression-<br>free survival | Alive: Free of progression | | • | | |
| _ | Total | | - | - | |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

Table 58. Time to PD (weeks) (Central assessment. ITT)

| | | Cohort A | | | Cohort B | | | tal | |
|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min- Max) | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |
| Time to | | | | | | | | _ | |
| PD | | | | | | | | | |
| (weeks) | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

Table 59. Follow-up time (weeks) (Central assessment. ITT)

| | | Cohort A | | | Cohort B | | | tal | |
|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) N | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |
| Follow- | | | | | | | | | |
| up time | | | | | | | | | |
| (weeks) | | | | | | | | | |
| 1: | | | | | Mann-W | hitneyU | | | tes |

<sup>2.7.4.</sup> PFS. CENTRAL ASSESSMENT. PP

Table 60. Progression-free survival at 12 and 24 weeks according to cohorts (Central

| _ | | ass | essment | . PP) | | • | |
|---|---|---|---|---|---|---|---|
| Progression-f | ree survival | N<br>events | N<br>patients<br>at risk | cumulati | timated<br>ve survival<br>atio | 95% CI | |
| | Cohort | | | | | | |
| at 12 weeks — | Α | | | | | | |
| at 12 weeks | Cohort | | | | | | _ |
| | В | | | | | | |
| | Cohort | | | | | | |
| ot 24 wooks — | Α | | | | | | |
| at 24 weeks — | Cohort | | | | | | _ |
| | В | | | | | | |
| | Strategy | N (%)<br>events | Median<br>(weeks) | Min-Max | Standard error | 95% CI | p-<br>value |
| Drawraaian — | Α | | | | • | | |
| Progression- free survival — | В | | | | | | _ |
| iree survival — | Total | | | | | | _ |
| | 1. Log ronk | toot | _ | | | | |

<sup>1:</sup> Log-rank test

#### Statistical analysis plan

Figure 4. Progression-free survival according to cohorts ( Central assessment. PP). Kaplan-Meier curve.

Table 61. Progression during follow-up (Central assessment. PP)

| | | Cohort A | Cohort B | Total | |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95% CI) | N (%,<br>95% CI) | — p-<br>value |
| | PD | | | | |
| Progression-<br>free survival | Alive: Free of progression | | | • | |
| | Total | | - | - | |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

Table 62. Time to PD (weeks) (Central assessment, PP)

| | | Cohort A | | | Cohort B | | | tal | |
|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min- Max) <sup>N</sup> | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |
| Time to PD | | | | | | | | _ | |
| (weeks) | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

Statistical analysis plan

#### **EFFICACY: ENDPOINT SECONDARY GLOBAL SURVIVAL (OS)** 2.8.

#### 2.8.1. OS. ITT

Table 63. Overall survival at 12 and 24 weeks according to cohorts (ITT)

| Overall survival | | N<br>events | N<br>patients<br>at risk | cumulati | timated<br>ve survival<br>atio | 95% CI | |
|---|---|---|---|---|---|---|---|
| | Cohort | | | | | | |
| at 12 | Α | | | | | | |
| weeks | Cohort | | | | | | |
| | В | | | | | | |
| | Cohort | | | | | | |
| at 24 | Α | | | | | | |
| weeks | Cohort | | | | | | |
| | В | | | | | | |
| | Strategy | N ( %)<br>events | Median<br>(weeks) | Min-Max | Standard<br>error | 95% CI | p-value |
| 0 | Α | | | | | | |
| Overall — | В | | | | | | |
| survival— | Total | | | | | | |
| | 1: Log | rank test | _ | | | | |

<sup>1:</sup> Log-rank test

Figure 5. Overall survival according to cohorts (ITT). Kaplan-Meier curve.

| | Table 64. Exitus o | luring follow-up | o and at 12 w | reeks (ITT) | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | |
| | | N (%, 95% CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | p-value |
| | Exitus | | | | |
| Overall | Live | | | | |
| survival | Loss Follow-up | | | | |
| | Total | | | | |
| | No | | | | |
| | Disease progression | · | | | |
| | Kidney failure | | | | |
| Reason<br>Exitus | Clinical deterioration | _ | | • | |
| | Post-surgical complications | == | | | |
| | Unknown | | | | |
| | Total Overall | | | • | |
| survival | Exitus | | | | |
| at 12 | Live | | | | |
| weeks | Total | | | • | |

<sup>1:</sup> Pearson Chi-square; 2: Fisher's exact test

Table 65. Time to exit (weeks) (ITT)

| | Cohort A | | | Cohort B | | | Tot | | |
|---|---|---|---|---|---|---|---|---|---|
| N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>1</sup> |

#### Statistical analysis plan

Exit time (weeks)

1: Mann-Whitney U test

#### 2.8.2. OS. PP

Table 66. Overall survival at 12 and 24 weeks according to cohorts (PP)

| Overal | Overall survival | | N patients<br>at risk | | ted cumulative<br>rival ratio | 95% CI | |
|---|---|---|---|---|---|---|---|
| at 12 | Cohort A | | | | | | |
| weeks | Cohort B | | | | | | |
| at 24 | Cohort A | | | | | | |
| weeks | Cohort B | | | | | | |
| | Strategy | N ( %)<br>events | Median<br>(weeks) | Min-Max | Standard error | 95% CI | p-value <sup>1</sup> |
| 0 | Α | | | | | | |
| Overall –<br>survival – | В | | | | | | |
| Sui VIVai — | Total | | | | | | |

1: Log-rank test

Figure 6. Overall survival according to cohorts (PP). Kaplan-Meier curve.

Table 67. Exitus during follow-up and at 12 weeks (PP)

| | | Cohort A | Cohort B | Total | |
|---|---|---|---|---|---|
| | | N (%, 95% CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | p-value |
| | Exitus | | | | |
| Over | rall Live | | | • | |
| surv | ival Loss Follow-up | | | • | |
| | Total | | | | |
| | No | | | | |
| | Disease | | | | - |
| | progression | | | | |
| | Kidney failure | | | | |
| Reas | son Clinical | <u> </u> | | • | |
| Exitu | us <u>deterioration</u> | | | | |
| | Post-surgical | | | | |
| | complications | | | | • |
| | Unknown | | | | |
| | Total Overall | | | | |
| surv | ival Exitus | | | | |
| at 12 | Live | | | · ——— | _ |
| weel | ks Total | | | • | - |

1: Pearson Chi-square; 2: Fisher's exact test
## Statistical analysis plan

Table 68. Time to exit (weeks) (PP)

| | Cohort A | | | Cohort B | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-<br>Max) | p-value <sup>2</sup> |
| Exit time (weeks) | • | | | | , | | | | , | |
| 1: | | | | | Mann-Whi | tney | | | | U-test |

Statistical analysis plan

#### 2.9. GMI: GROWTH MODULATION INDEX

Following the definition in the protocol, the GMI will be calculated as "the ratio between time to progression with pazopanib (TTPp) divided by time to progression with the previous line of treatment (TTPp-1)".

The time to PD with pazopanib is presented in the section EFFICIENCY: MAIN ENDPOINT and the duration of the previous chemotherapy until relapse is presented in Table 30. Number of cycles and duration of the previous chemotherapy.

Table 69. Growth modulation index (GMI) (ITT)

| | | Cohort A | | | Cohort B | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max) | value <sup>1</sup> |
| Growth modulation | | | | | | | | | | |
| index (GMI) | | | | | | | | | | |

<sup>1:</sup> Mann-Whitney U test

Table 70. Categorized GMI (ITT)

| | | Cohort A | Cohort B | Total | p-value |
|-------------|--------|----------|----------|-------|---------|
| | _ | N (%) | N (%) | N (%) | |
| | <1 | | | | |
| GMI | 1-1.33 | | | | |
| categorized | > 1.33 | | | | |
| | Total | | | | |

1: Chi-square; 2: Fisher's exact test

| Table 71. Growth modulation index (GMI) (PP) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Co | hort A | | Co | hort B | | Total | p-<br>value <sup>1</sup> |
| | N Mean<br>(SD) | Median<br>(Min-Max) | N | Mean<br>(SD) | Median<br>(Min-Max ) | N Mean<br>(SD) | Median<br>(Min-Max) | |

| Growth | |
|------------|-------|
| modulation | index |
| (GMI) | |

<sup>1:</sup> Mann-Whitney U test

Table 72. Categorized GMI (PP)

| | | | rategerizea e iii (i i ) | | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | p-value |
| | | N (%) | N ( %) | N (%) | |
| | <1 | | | | |
| CMI | 1-1.33 | | | | |
| GMI<br>categorized | > 1.33<br>Total | | | | |
| categorized | Total | | | | |
| | 4 0 | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

#### 2.10. ECOG EVOLUTION

Table 73. ECOG evolution during treatment (ITT)

| | Table 73. ECOG | | | Τ) | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | |
| | | N (%) | N (%) | N (%) | p-value |
| Performance | 0 | | | | |
| Status ECOG | 1 | | | | |
| (baseline) | Total | | | | |
| Performance _ | 0 | | | | |
| ECOG Status | 1 | | | | |
| Day 1 | Total | | | | |
| Df | 0 | | | | |
| Performance — Status ECOG — | 1 | | | | |
| Week 1 — | 2 | | | | |
| Week i — | Total | | | | |
| Performance | 0 | | | | |
| Status ECOG | 1 | | | | |
| Week 3 | Total | | | | |
| | 0 | | | | |
| Performance - | 1 | | | | |
| Status ECOG — Week 5 — | 2 | | | | |
| week 5 — | Total | | | | |
| | 0 | | | | |
| Performance — | 1 | | | | |
| Status ECOG – Week 7 – | 2 | | | | |
| Week / | Total | | | | |
| | 0 | | | | |
| Performance — | 1 | | | | |
| Status ECOG – Week 9 – | 2 | | | | |
| week 5 — | Total | | | | |
| Performance | 0 | | | | |
| Status ECOG | 1 | | | | |
| Week 12 | Total | | | | |
| | Basal vs. day 1 | | | | |
| | Basal vs. week 1 | | | | |
| | Basal vs. week 3 | | | | |
| p-value <sup>3</sup> | Basal vs. week 5 | | | | |
| · | Basal vs. week 7 | | | | |
| | Basal vs. week 9 | | | | _ |
| _ | Basal vs. week 12 | _ | | | |
| 1. Dooroon's Chi o | guara: 2: Fishar's avast tool | t. O. Manainal hans | | | <del></del> |

<sup>1:</sup> Pearson's Chi-square; 2: Fisher's exact test; 3: Marginal homogeneity test

#### 2.11. SAFETY: SAEs AND TOXICITIES

Following the criteria established in the protocol, "Any patient included in the study and who has received at least a single dose of study medication will be evaluable for toxicity analyzes."

#### Statistical analysis plan

AES and Toxicities Table 74. All monitoring

| | | CohortA | Cohort B | Total | – p-value |
|---------------------------|-------|---------|----------|-------|-------------|
| | | N (%) | N (%) | N (%) | – p-value |
| A <b>-</b> | Yes | | • | | |
| AE - | Total | | | | <del></del> |
| toxicity<br>(related) | No | | - | | |
| | Yes | | - | | |
| | Total | • | • | | |
| | No | | - | | |
| ≥3 AE grade | Yes | | | | |
| - | Total | | - | | |
| tovioity grada | No | • | • | | |
| toxicity grade - | Yes | | | | |
| ≥3 (related) <sup>-</sup> | Total | | - | | |
| SAE (at least | No | • | • | | |
| one per | Yes | • | • | | |
| patient) <sup>3</sup> | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test; 3: patients could present more than one SAE

Table 75. AEs and Toxicities with start date prior to treatment

| Tubic 70 | ,, , L=3 und | TOXIOICIOS WITH | Start date prior | to troutino | |
|---|---|---|---|---|---|
| | | Cohort A | Cohort B | Total | — p-value |
| | | N (%) | N (%) | N (%) | — p-value |
| • | No | • | • | | |
| AE | Yes | • | • | | |
| _ | Total | | | | |
| AE grade ≥ 3 | No | • | • | | |
| | Total | • | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Table 76. AEs and Toxicities during treatment

| | Cohort A | Cohort B | Total | — p-value |
|---|---|---|---|---|
| | N (%) | N (%) | N (%) | — p-value |
| Yes | • | • | | |
| Total | | | | |
| No | • | | | |
| Yes | • | | | |
| Total | • | | | |
| No | • | | | |
| Yes | | | | <del></del> |
| Total | • | | | <del></del> |
| No | • | | | |
| Yes | | | | |
| Total | • | • | | <del></del> |
| | Total No Yes Total No Yes Total No Yes Total No | N (%) Yes Total No Yes Total No Yes Total No Yes Total No Yes | N (%) N (%) Yes Total No Yes Total No Yes Total No Yes Total No Yes | N (%) N (%) N (%) Yes Total No Yes Total No Yes Total No Yes Total No Yes |

**Table 77. ESA and Toxicities after treatment** 

| | | Cohort A | Cohort B | Total | — p-value |
|---|---|---|---|---|---|
| | | N (%) | N (%) | N (%) | — p-value |
| | No | • | · | | |
| AE | Yes | • | - | | |
| | Total | | | | |

#### Statistical analysis plan

| Toxicity (related) | No | | · |
|---|---|---|---|
| | Yes | · | |
| | Total | , | |
| AE grade ≥3 | No | , | |
| | Yes | | <u> </u> |
| _ | Total | , | |
| Toxicity grade | No | , | |
| ≥3<br>(related) | Total | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Table 78. AE and Toxicities with no known date

| | | Cohort A | Cohort B | Total | — p-value |
|----------------|-------|----------|----------|-------|-------------|
| | | N (%) | N (%) | N (%) | — p-value |
| | No | • | • | | |
| AE | Yes | - | | | |
| _ | Total | | | | <del></del> |
| Tarrialtar | No | | | | |
| Toxicity - | Yes | - | | | |
| (related) – | Total | - | | | |
| | No | | | | · |
| AE grade ≥3 | Yes | - | | | |
| _ | Total | - | | | |
| Toxicity grade | No | | | | |
| ≥3 (related) | Total | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

The frequencies of all toxicities with grade ≥3 are presented below.

Table 79. Frequencies of AEs grade ≥ 3

| | Cohort A | Cohort B | Total |
|--------------------------------------------|----------|----------|-------|
| | N (%) | N (%) | N (%) |
| Abscess of tumor mass - Grade 3 | | | |
| ALT increased - Grade 3 | | | |
| Anemia - Grade 3 | | | |
| Ascites - Grade 3 | | | |
| AST increased - Grade 3 | | | |
| Asthenia - Grade 3 | | | |
| Back pain - Grade 3 | | | |
| Bilirubin increased - Grade 3 | | | |
| Cardiac dysrhythmia / chest pain - Grade 3 | | | |
| Diarrhea - Grade 3 | | | |
| Fatigue - Grade 3 | | | |
| Femur fracture - Grade 3 | | | |
| Gastrointestinal bleeding - Grade 5 | | | |
| General Status deterioration - Grade 5 | | | |
| Ggt increased worsening - Grade 3 | | | |
| Hypertension - Grade 3 | | | |
| Hyporexia - Grade 3 | | | |
| Muscle weakness - Grade 3 | | | |
| Myocardial infarction - Grade 3 | | | |
| Nausea - Grade 3 | | | |
| Neutropenia - Grade 3 | | | |

#### Statistical analysis plan

| Pain - Grade 3 |
|---------------------|
| Toothache - Grade 3 |
| Vomiting - Grade 3 |

The frequencies of all (related) treatment toxicities with grade ≥3.

Table 80. Frequencies of (related) toxicities grade ≥ 3

| | Cohort A | Cohort B | Total |
|---------------------------------|----------|----------|-------|
| | N (%) | N (%) | N (%) |
| ALT increased - Grade 3 | | | |
| AST increased - Grade 3 | | | |
| Asthenia - Grade 3 | | | |
| Bilirubin increased - Grade 3 | | | |
| Diarrhea - Grade 3 | | | |
| Hypertension - Grade 3 | | | |
| Muscle weakness - Grade 3 | | | |
| Myocardial infarction - Grade 3 | | | |
| Nausea - Grade 3 | | | |
| Neutropenia - Grade 3 | | | |
| Vomiting - Grade 3 | | | |
| | | · | |

## Statistical analysis plan

All reported SAEs are listed below, by cohort.

| Table 81. | List of | of all | SAEs | reported |
|-----------|---------|--------|------|----------|
|-----------|---------|--------|------|----------|

| Coho<br>rt ID | Hospital | Sex | Toxicity | Paz \ 0. | When the AE is presented | StartT<br>X | dateE<br>nd<br>date<br>AE | Result | Continue<br>d | SA SAE<br>E solution |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | · | |
| | | | | | | * | | | | |

In APPENDIX II: LISTED ALL TOXICITIES RELATED

Statistical analysis plan

#### 3. APPENDIX I: EFFICACY ACCORDING TO GMI

#### 3.1. ENDPOINT MAIN ACCORDING TO GMI

In the sections presented below, the possible relationship between the main efficacy variables and the categorized GIM variables is analyzed: <1, 1-1.33 and> 3 (see Table 69. Growth modulation index (GMI) (ITT) and Table 71. Modulation index Growth (GMI) (PP).

# 3.1.1. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. ITT

The tables below show the response to treatment at 6 and 12 weeks, based on *local assessments* of the TACs based on the categorized GMI variable: <1, 1-1.33 and> 3.

Table 82. Response to treatment according to GMI: Local assessment at 6 and 12 weeks

| | | | ized | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | |
| | | N (%, 95%<br>CI) | %N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95% CI) | p-value |
| Clinical benefit at | No<br>(PD) | | | , | | |
| week 6 (CR, PR or SD) local | Yes | | | | | |
| | Total | | <del>.</del> | | | |
| Clinical benefit at | No | | | | | |
| | (PD) | | | | | |
| week 12 (CR, PR or | Yes | • | • | | | |
| SD) local | Total | • | • | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

# 3.1.2. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. PP

Table 83. Response to treatment according to GMI: Local evaluations at 6 and 12 weeks PP

| | | <1 | 1-1.33 | > 1.33 | Total | |
|---|---|---|---|---|---|---|
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (% ,<br>95% CI) | N (%, 95% CI) | p-value |
| Clinical benefit at | No<br>(PE) | | | | | |
| week 6 (CR, PR or -<br>SD) local | Yes<br>Total | | | | | |
| Clinical benefit at | No<br>(PE) | • | | | | |
| week 12 (CR, PR or<br>SD) local | Yes<br>Total | | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

# 3.1.3. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. ITT. IN EACH COHORT

The tables shown below show the **response to treatment at 6 and 12 weeks**, in the **ITT population**, based on **local assessments** of TACs based on the categorized GMI variable: <1, 1-1.33 and> 3, separated according to each cohort.

Table 84. Response to treatment according to GMI: local assessments at 6 and 12 weeks ITT. Cohort A

| | | <1 | 1-1.33 | > 1.33 | Total | |
|---|---|---|---|---|---|---|
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95% CI) | p-value |
| Clinical benefit at | No<br>(PD) | | | | | |
| week 6 (CR, PR or SD) local | Yes | | | | | |
| SD) local | Total | | | • | | |
| Clinical benefit at | No<br>(PD) | | | | | |
| week 12 (CR, PR or | Yes | | | | | |
| SD) local | Total | | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Table 85. Response to treatment according to GMI: Local assessments at 6 and 12 weeks ITT. Cohort B

| | | | GMI categorized | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | |
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95% CI) | p-value |
| Clinical benefit at | No<br>(PD) | | | | | |
| week 6 (CR, PR or<br>SD) local | Yes | | | | | <del>_</del> |
| <u> </u> | Total | | | | | |
| Clinical benefit at | No<br>(PD) | | | | | |
| week 12 (CR, PR or | Yes | | | | | <u> </u> |
| SD) local | Total | • | | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

# 3.1.4. RESPONSE LOCAL ASSESSMENTS AND ACCORDING TO GMI. PP. IN EACH COHORT

The tables shown below show the **response to treatment at 6 and 12 weeks,** in the **PP population,** based on **local assessments** of TACs based on the categorized GMI variable: <1, 1-1.33 and> 3, separated according to each cohort.

Table 86. Response to treatment according to GMI: Local evaluations at 6 and 12 weeks PP. Cohort A

| | | GMI categorized | | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | |
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95% CI) | p-value |
| Clinical benefit a week 6 (CR, PR or | No<br>(PD) | | | | | |

#### Statistical analysis plan

| SD) local | Yes | _ |
|---------------------------------|------------|---|
| | Total | _ |
| Clinical benefit at | No<br>(PD) | _ |
| week 12 (CR, PR or<br>SD) local | Yes | _ |
| SD) local | Total | _ |

1: Chi-square; 2: Fisher's exact test

Table 87. Response to treatment according to GMI: Local assessments at 6 and 12 weeks PP. Cohort B

| | | <1 | 1-1.33 | > 1.33 | Total | |
|---|---|---|---|---|---|---|
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95% CI) | p-value |
| Clinical benefit a | No<br>(PD) | | , | | | |
| week 6 (CR, PR or SD) local | Yes<br>Total | | | | | |
| Clinical benefit at | No<br>(PD) | | | | | |
| week 12 (CR, PR or<br>SD) local | Yes | | | | | |
| 3D) IOCAI | Total | | | | | |
| 1: | | Chi-square; | | 2: | Fisher | exact |

Statistical analysis plan

#### 3.2. SECONDARY ENDPOINT PFS ACCORDING TO GMI

#### 3.2.1. PFS ACCORDING TO GMI. LOCAL ASSESSMENT

Figure 7. PFS according to GMI (Local Assessment. ITT). Kaplan-Meier curve.

Table 88. PFS according to GMI (Local assessment. ITT)

| | ruble 66: 11 6 decording to Gilli (200di doscosilient: 111) | | | | | |
|---|---|---|---|---|---|---|
| | GMI | N (%)<br>events | Median<br>(weeks) | Standard error | 95% CI | p-value <sup>1</sup> |
| | <1 | | | | | |
| PFS | 1-1.33 | | | | | |
| PFS | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

Figure 8. PFS according to GMI (Local Assessment. PP). Kaplan-Meier curve.

Table 89. PFS according to GMI (Local assessment. PP)

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| DEC | 1-1.33 | | | | | |
| PFS | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

# 3.2.2. PFS ACCORDING TO GMI . LOCAL ASSESSMENT. IN COHORT A

Figure 9. PFS according to GMI (local assessment. ITT). Kaplan-Meier curve. Cohort A

Table 90. PFS according to GMI (local assessment. ITT) Cohort A

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| DEC | 1-1.33 | | | | | |
| PFS | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Test of Log- rank

Figure 10. PFS according to GMI (Local assessment. PP). Kaplan-Meier curve. Cohort A

Table 91. PFS according to GMI (local assessment. PP) Cohort A

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| PFS | 1-1.33 | | | | | |
| PFS | > 1.33 | | | | | |
| | Overall | | | | | |

#### Statistical analysis plan

1: Log Test- rank

# 3.2.3. PFS ACCORDING TO GMI. LOCAL ASSESSMENT. IN COHORT B

Figure 11. PFS according to GMI (local assessment. ITT). Kaplan-Meier curve. Cohort B

Table 92. PFS according to GMI (local assessment. ITT) Cohort B

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| PFS | 1-1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

Figure 12. PFS according to GMI (Local assessment. PP). Kaplan-Meier curve. Cohort B

Table 93. PFS according to GMI (local assessment. PP) Cohort B

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| PFS | 1-1.33 | | | | | <u> </u> |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

#### 3.3. SECONDARY ENDPOINT OS ACCORDING TO GMI

#### 3.3.1. OS ACCORDING TO GM.

Figure 13. OS according to GMI (ITT). Kaplan-Meier curve.

Table 94. OS according to GMI (ITT)

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| 00 | 1-1.33 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

Statistical analysis plan

Figure 14. OS according to GMI (PP). Kaplan-Meier curve.

Table 95. OS according to GMI (PP)

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | _ |
| 00 | 1-1.33 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

#### 3.3.2. OS ACCORDING TO GMI. IN COHORT A

Figure 15. OS according to GMI (ITT). Kaplan-Meier curve. Cohort A

Table 96. OS according to GMI (ITT) Cohort A

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| 00 | 1-1.33 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

Figure 16 OS according to GMI (PP). Kaplan-Meier curve. Cohort A

Table 97. OS according to GMI (PP) Cohort A

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| 00 | 1-1.33 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

### 3.3.3. OS ACCORDING GMI. IN COHORT B

Figure 17. OS according to GMI (ITT). Kaplan-Meier curve. Cohort B

Table 98. OS according to GMI (ITT) Cohort B

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

<sup>1:</sup> Log-rank test

#### Statistical analysis plan

Figure 18. OS according GMI (PP). Kaplan-Meier curve. Cohort B

Table 99. OS according to GMI (PP) Cohort B

| | GMI | N (%)<br>events | Median<br>(weeks) | Standard<br>error | 95% CI | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | <1 | | | | | |
| os | > 1.33 | | | | | |
| | Overall | | | | | |

1: Log-rank

Statistical analysis plan

### 3.4. ECOG test (BASAL) ACCORDING GMI

#### 3.4.1. ECOG BASAL ACCORDING TO GMI. ITT

The following tables analyze the possible relationship between the variables ECOG baseline and categorized GMI: <1, 1-1.33 and> 3.

Table 100. Baseline ECOG according to GMI (ITT)

| | | GMI categorized | | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | |
| | | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (%, 95%<br>CI) | N (% , 95% CI) | p-value |
| D | 0 | · | • | | | |
| Performance<br>status | 1 | | | | | |
| Siaius | Total | | | | | |

<sup>1:</sup> Chi-square; 2: Fisher exact test

#### 3.4.2. ECOG BASAL ACCORDING TO GMI. PP

Table 101. Baseline ECOG according to GMI (PP)

| | | <1 | 1-1.33 | > 1.33 | Total | |
|---|---|---|---|---|---|---|
| | | N (%,<br>95% CI) | N (%, 95%<br>CI) | N (%,<br>95% CI) | N ( %, 95% CI) | p-value |
| Doufousson | 0 | • | • | • | | |
| Performance status | 1 | | | | | <del></del> |
| Status | Total | • | • | | | <del></del> |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

#### 3.5. GRADE FNCLCC (BASAL) ACCORDING TO GMI

# 3.5.1. GRADE FNCLCC BASAL ACCORDING TO GMI. ITT

The following tables analyze the possible relationship between the variables grade FNCLCC baseline and categorized GMI: <1, 1-1.33 and> 3.

Table 102. GRADE FNCLCC baseline according to GMI (ITT)

| | | GMI categorized | | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | р- |
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | N ( %, 95% CI) | value |
| - | 1 | • | | | • | |
| GRADE | 2 | | | | | -<br>-0.017 <sup>2</sup> |
| FNCLCC | 3 | | | | | 0.017 |
| | Total | • | | | • | <u> </u> |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

Statistical analysis plan

## 3.5.2. GRADE FNCLCC BASAL ACCORDING TO GMI. PP

Table 103. GRADE FNCLCC baseline according to GMI (PP)

| | | GMI categorized | | | | |
|---|---|---|---|---|---|---|
| | | <1 | 1-1.33 | > 1.33 | Total | p- |
| | | N (%, 95% CI) | N (%, 95% CI) | N (%, 95% CI) | N ( %, 95% CI) | value |
| | 1 | | | | | |
| GRADE | 2 | · | | | • | _ |
| FNCLCC | 3 | - | | | • | = |
| | Total | | | | | |
| | 4. 01-1 | ro. 2. Fisher's ever | 444 | | | |

<sup>1:</sup> Chi-square; 2: Fisher's exact test

## 4. ANNEX II: LISTING OF ALL RELATED

TOXICITIES All the related toxicities collected in the database are listed below, by cohort.

| | | | | Table 104. List of all related toxicities | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort ID | Hospital | Sex | Toxicity | Relati<br>ve.<br>Pazo. | When the AE is presented | StartT<br>X | dateSt<br>art | date<br>AE<br>End<br>date<br>AE | Result | Continuo<br>us | SA SAE<br>E solution |
| | | | | • | | | | | | • | |
| <del></del> | | | | • | | | | | | * | |
| | | | | | | | | | | * | |
| | | | | • | | | | | | * | |
| | | | | | | | | - | | | |